CLINICAL TRIAL: NCT03455725
Title: Randomized Controlled Pivotal Trial of Autologous Bone Marrow Cells Using the CardiAMP Cell Therapy System in Patients With Refractory Angina Pectoris and Chronic Myocardial Ischemia (CardiAMP CMI Trial)
Brief Title: CardiAMP Cell Therapy Chronic Myocardial Ischemia Trial
Acronym: CardiAMP-CMI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioCardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04747 (CLIN)
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Refractory Angina; Chronic Myocardial Ischemia
Keywords: Cardiovascular Stem Cell Therapy; Bone Marrow Mononuclear Stem Cells; Intramyocardial Injection
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, 2:1 randomized (Treatment vs Sham Control), blinded trial comparing 2 paralel groups of patients with CMI treated with CardiAMP cell therapy system vs sham treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple-blinded, placebo-controlled study. Patients, investigators, the CRO, core labs and the sponsor will be blinded for individual treatment adjudication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CardiAMP cell therapy system (Active Comparator): Roll-in phase:
  Up to 10 subjects with refractory chronic myocardial ischemia CCS class III-IV will be treated in an unblinded, uncontrolled roll-in phase.
  In the subsequent randomized phase:
  Up to 333 subjects with refractory chronic myocardial ischemia CCS class III-IV will be randomized. Up to 222 Subjects will be randomized to treatment with the CardiAMP cell therapy system.
  Interventions: Device: CardiAMP Cell Therapy System
- Sham procedure control (Sham Comparator): Randomized phase:
  Up to 333 subjects with refractory chronic myocardial ischemia CCS class III-IV will be randomized. Up to 111 subjects will be treated with a Sham Treatment (no introduction of trans endocardial delivery catheter and no administration of autologous cells)
  Interventions: Other: Sham Treatment

INTERVENTIONS:
Device: CardiAMP Cell Therapy System — The CardiAMP Cell Therapy system consists of the CardiAMP Potency Assay, the Helix/Morph intramyocardial delivery catheter system, and the CardiAMP Cell Separator. The system allows the investigator to identify patients with a high chance to respond to im autologous stem cell therapy (using the CardiAMP Cell Potency Assay), to isolate the stem cells from a bone marrow harvest at the point of care (using the CardiAMP CS system), and to percutaneously inject the autologous cells into the myocardium using the Helix/Morph delivery catheters.
  Arms: CardiAMP cell therapy system
Other: Sham Treatment — Patients will receive sham bone marrow procedure and a ventriculogram. A scripted sham percutaneous procedure will be performed
  Arms: Sham procedure control

SUMMARY:
Prospective, multi-center, 2:1 randomized (Treatment : Sham Control), sham-controlled, double-blinded trial to compare treatment using the CardiAMP cell therapy system to sham treatment

Treatment Group:

Subjects treated with aBMC using the CardiAMP cell therapy system

Sham Control Group:

Subjects treated with a Sham Treatment (no introduction of the Helix transendocardial delivery catheter, no administration of aBMC)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 21 to 80 years of age
2. Canadian Cardiovascular Society (CCS) class III or IV chronic refractory angina.
3. Lack of control of angina symptoms despite maximum tolerated doses of anti-angina drugs.
4. Evidence of inducible myocardial ischemia on baseline stress testing
5. Obstructive coronary disease unsuitable for conventional revascularization
6. Experience angina episodes at a minimum of 7 angina episodes per week (during a 4-week screening period).
7. Able to complete an exercise tolerance test on the treadmill
8. Left ventricular ejection fraction of greater than or equal to 40% as measured by echocardiography.
9. Qualification of a pre-procedure screening of bone-marrow aspiration

Exclusion Criteria

Other cardiac or vascular system or other health-related criteria which may be seen in a patient's history and physical examination.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Total Exercise Time on the treadmill using the Modified Bruce Protocol | Baseline and 6 months visit
  A superiority analysis with regards to change from Baseline in Total Exercise Time at the 6 months follow-up visit (using a Modified Bruce Protocol).

SECONDARY OUTCOMES:
Safety: overall survival at 6 months follow-up | at 6 months follow-up
  A non-inferiority analysis of overall survival at 6-months will be made comparing the Treatment group to the Sham Control group using a non-inferiority margin of 10%.
Safety: Total Major adverse cardiac events (MACE) at 6 months follow-up | from randomisation to 6 months follow-up
  A non-inferiority analysis with regard to Total Major Adverse Cardiac Events (MACE: defined as death, cardiac hospitalization, non-fatal myocardial infarction and stroke) at 12 month follow-up, as adjudicated by an independent clinical endpoint classification (CEC) committee with 10% margin.
Efficacy: Change from baseline in Total Exercise Time at 6 months follow-up | Baseline and at 6 months follow-up
  Superiority analysis with regards to change from baseline in Total Exercise Time on Exercise Tolerance Test (ETT) at 6 Month Follow-up Visit. Baseline (BL) is the average of (at least) two total exercise times measured during the screening period.
Efficacy: Change of angina frequency (per week) at 12 months follow-up | Baseline and at 12 months follow-up
  Superiority analysis with regards to change in angina frequency (episodes per week) at 12 month follow-up Visit versus baseline angina frequency (per week).
  Participants self-reported angina episodes utilizing an electronic diary for 4 weeks at baseline (screening period) and in the 4 weeks before the 12-month follow-up visits.
Efficacy: Change of Angina Frequency (per week) at 6 months follow-up | Baseline and at 6 months follow-up
  Superiority analysis with regards to change in angina frequency at 6 month follow-up visit versus baseline (expressed as angina frequency per week).
  Participants self-reported angina episodes utilizing an electronic diary for 4 weeks at baseline and in the 4 weeks before the 6-month follow-up visits.
Safety: Total Major adverse cardiac events (MACE) at 12 months follow-up | From randomisation to 12 month follow-up
  Superiority analysis with regards to incidence of MACE from Randomization until the end of the 24 month follow-up period
Efficacy: Percentage of patients with at least 1 Serious Adverse Event (SAE) | From randomization to 12 Months follow-up
  Superiority analysis with regards to percentage of participants with at least one SAE. From randomization until the end of the 12 month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Amish Raval, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Wisconsin Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: company website — http://biocardia.com